CLINICAL TRIAL: NCT02225925
Title: Phase II Study of Dynamic Intraoperative Dosimetry for Prostate Brachytherapy Using Registered Fluoroscopy and Ultrasound
Brief Title: Intraoperative Dosimetry for Prostate Brachytherapy Using Fluoroscopy and Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J13164; NA_00091766 (Other: JHMIRB)
Record Dates: First submitted 2014-04-08; First posted 2014-08-26 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dynamic dosimetry brachytherapy (Experimental): Cohort treated with dynamic dosimetry brachytherapy
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy

SUMMARY:
The purpose of this study is to assess the performance of a system of intraoperative dynamic dosimetry during prostate seed implantation (brachytherapy) including its new elements, to evaluate and refine technical methods of using the system, as well as confirm its performance and accuracy.

DETAILED DESCRIPTION:
The use of brachytherapy or implantation of radioactive sources into the prostate for adenocarcinoma has advantages over external beam radiation in that a very high dose can be delivered to the tumor while limiting the doses to the surrounding normal tissue (i.e., bowel and bladder). It is established that outcomes after treatment with brachytherapy are related to the technical quality of source placement within the gland. Accurate placement of the radioactive sources with achievement of optimum dose distributions within the prostate is key to the success of brachytherapy with regard to both killing tumor as well as minimizing toxicity.

Due to factors such as deformations of the prostate during needle insertion, needle deviation from intended path during insertion, prostatic edema from needle trauma, and relaxation of tissues as well as source migration after needle removal, the actual source positions upon completion of the procedure may fail to accurately match their intended placement, resulting in variations from the idealized dosimetric plan.

One way to overcome this complex problem is to have the capability of visualizing the sources once they are in the prostate and then continuously updating the dosimetric plan in real time. To this end, we have developed a mechanism whereby ultrasound and fluoroscopy are quantitatively integrated to allow for real-time visualization of source positions intraoperatively. A prior Phase I study performed by this group evaluated a prototype version of this mechanism, resulting in the successful treatment of 6 patients with true intraoperative dynamic dosimetry. Dosimetric outcomes within this cohort of patients was excellent, and the intraoperative doses predicted by the system more accurate than that predicted by the current standard method (ultrasound-based dosimetry).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, localized adenocarcinoma of the prostate
* Clinical stages T1b - T3a
* The patient has decided to undergo brachytherapy (or brachytherapy plus external beam radiation) as a treatment modality for his prostate cancer
* Karnofsky Performance Status > 60
* Prostate volume by transrectal ultrasound (TRUS) < 55 cc
* International Prostate symptom score (IPSS) 20 or less
* Ability to have Magnetic resonance imaging as part of post-implant assessment
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Stage T3b or greater disease.
* Prior history of pelvic radiation therapy
* Significant obstructive symptoms (IPSS greater than 20)
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow up.
* Implanted device or apparatus which obstruct visibility of the implanted sources on fluoroscopy
* Metallic implants, claustrophobia not amenable to medication, or known contraindications to undergoing MR scanning

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 45 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Song, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (1):
- The SKCCC at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dynamic Dosimetry Brachytherapy
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 29
Age, Continuous [Mean (Full Range); unit: years] | 68 [55 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: Additional procedure time with the registered ultrasound and fluoroscopy system (RUF) in the intra-operative setting for implantation procedure
Time Frame: at time of implantation procedure
Measure: Mean (Full Range); unit: minutes
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 45
minutes | 30 [14 to 45]

2. Secondary Outcome: Seed Reconstruction From Intra-operative Fluoroscopy
Description: Number of patients with all seeds reconstructed from fluoroscopy
Time Frame: up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 45
Participants | 45

3. Secondary Outcome: Number of Participants With Seed Reconstruction Utilizing RUF Versus CT / Magnetic Resonance Imaging (MRI) Reconstruction
Description: Number of participants with seed reconstruction with RUF versus CT fused with MRI doses for Prostate D90 (dose received by 90% of prostate)
Time Frame: 30 days post-treatment
Population: Data was not collected to assess this outcome measure
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Impact of RUF System on Dosimetric Outcomes of Seed Placement as Assessed by Number of Patients With Prostate V100 of 95% or Greater
Description: Number of patients with prostate V100 (the percent of the postimplant MR/CT-based prostate volume that received at least 100% of dose) of 95% or greater
Time Frame: 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 45
Participants | 44

5. Secondary Outcome: Mean Difference in D90 Between Intra-operative RUF and Standard CT/MRI Based Dosimetry
Description: Mean difference of D90 (% of prescribed dose) between intra-operative RUF and standard CT/MRI based dosimetry
Time Frame: Treatment - 30 days
Measure: Mean (95% Confidence Interval); unit: percentage of prescribed dose
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 45
percentage of prescribed dose | 8 [6 to 10]

6. Secondary Outcome: Dosimetric Accuracy Comparison Between Pre and Post Ultrasound (US) Implantation Prostate Edema
Time Frame: Treatment - 30 days
Population: Data was not collected to assess this outcome measure
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Quality of Life (QoL) Assessments
Description: Change in Quality of Life measures based on International Prostate Symptom Score (range 0-35, higher score reflects lower quality of life), Sexual Health Inventory Score (1-25, lower score reflects lower quality of life), Epic-26 Bowel score (0-100, lower score reflects lower quality of life)
Time Frame: baseline, 30 days post-implant, semiannually post treatment until year 2 and then annually until year 5
Population: Data was not collected to assess this outcome measure
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 0

8. Secondary Outcome: Prostate Specific Antigen (PSA) Outcomes
Description: PSA biochemical failure-free survival at last follow-up visit
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Dosimetry Brachytherapy
Number analyzed (Participants) | 45
Participants | 45

ADVERSE EVENTS:
Time Frame: AEs were assessed for serious (Grade 3+) and/or unexpected events (those not expected/known risks of treatment); during treatment and up to 60 days after treatment.
Description: This is a research trial that is studying the feasibility and practicability of a new treatment planning system for patients who undergo brachytherapy. There are no expected adverse events associated with this trial, however, the research team will conduct post-follow-ups on all patients enrolled in this trial to report any adverse events (AEs) that are either unexpected or serious.
  No AEs or mortality were reported during this period.
Arm/Group | Dynamic Dosimetry Brachytherapy
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No